CLINICAL TRIAL: NCT02474173
Title: Phase 1b Study of HSP90 Inhibitor, AT13387 (Onalespib) in Combination With Paclitaxel in Patients With Advanced, Triple Negative Breast Cancer
Brief Title: Onalespib and Paclitaxel in Treating Patients With Advanced Triple Negative Breast Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Drug supply issues
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2015-00866; NCI-2015-00866 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); OSU 15149; 9876 (Other: Ohio State University Comprehensive Cancer Center LAO); 9876 (Other: CTEP); UM1CA186712 (NIH)
Record Dates: First submitted 2015-06-15; First posted 2015-06-17 (Estimated); Last update posted 2022-11-04 (Actual); Status verified 2022-11

CONDITIONS: Advanced Breast Carcinoma; Metastatic Breast Carcinoma; Stage III Breast Cancer AJCC v7; Stage IIIA Breast Cancer AJCC v7; Stage IIIB Breast Cancer AJCC v7; Stage IIIC Breast Cancer AJCC v7; Stage IV Breast Cancer AJCC v6 and v7; Triple-Negative Breast Carcinoma
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms | interventions — (2,4-dihydroxy-5-isopropylphenyl)-(5-(4-methylpiperazin-1-ylmethyl)-1,3-dihydroisoindol-2-yl)methanone; Paclitaxel; Taxes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (onalespib, paclitaxel) (Experimental): SAFETY RUN-IN: Patients receive onalespib IV over approximately 1 hour on day -7.
  TREATMENT: Patients receive paclitaxel IV over 60 minutes on day 1, 8, and 15. Patients also receive onalespib IV over 1 hour beginning on days 8 and 15 of cycle 1 and on days 1, 8, and 15 of subsequent cycles. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Drug: Onalespib; Drug: Paclitaxel; Other: Pharmacological Study

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Onalespib — Given IV
  Other Names: AT 13387; AT-13387; AT13387
Drug: Paclitaxel — Given IV
  Other Names: Anzatax; Asotax; Bristaxol; Praxel; Taxol; Taxol Konzentrat
Other: Pharmacological Study — Correlative studies

SUMMARY:
This phase Ib trial studies the side effects and best dose onalespib when given together with paclitaxel in treating patients with triple negative breast cancer that has spread to other places in the body and usually cannot be cured or controlled with treatment (advanced). Onalespib works by blocking proper processing of proteins that are important for cancer growth. This results in inability of these proteins to work properly. Paclitaxel kills breast cancer cells by interfering with their ability to divide. Giving onalespib together with paclitaxel may be better than giving either one alone in treating patients with breast cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the recommended phase 2 dose (RP2D) of onalespib (AT13387) in combination with paclitaxel in patients with advanced triple negative breast cancer (TNBC).

II. To determine the toxicity profile (based on Common Terminology Criteria for Adverse Events [CTCAE] version [v.]5.0) of the combination of AT13387 in combination with paclitaxel in patients with advanced TNBC.

SECONDARY OBJECTIVES:

I. To determine the effect of AT13387 on pharmacokinetics of paclitaxel in the study patient population.

II. To determine the effect of paclitaxel on pharmacokinetics of AT13387 in the study patient population.

III. To observe anti-tumor activity determining the overall response rate (partial response + complete response), response duration and progression-free survival.

OUTLINE: This is a dose-escalation study of onalespib.

SAFETY RUN-IN: Patients receive onalespib intravenously (IV) over 1 hour on day -7.

TREATMENT: Patients receive paclitaxel IV over 60 minutes on day 1, 8, and 15. Patients also receive onalespib IV over 1 hour beginning on days 8 and 15 of cycle 1 and on days 1, 8, and 15 of subsequent cycles. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed measurable or unmeasurable advanced or metastatic breast cancer for which standard curative measures do not exist or are no longer effective

  * Measurable disease is defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for non-nodal lesions and short axis for nodal lesions) as >= 20 mm (>= 2 cm) with conventional techniques or as >= 10 mm (>= 1 cm) with spiral computed tomography (CT) scan, magnetic resonance imaging (MRI), or calipers by clinical exam
* Primary and/or metastatic breast tumor must be negative for over-expression of estrogen and progesterone receptors; patients with weak estrogen receptor and/or progesterone receptor expression (< 10% on immunohistochemistry [IHC]) will be eligible
* Primary and/or metastatic breast tumor must be negative for human epidermal growth factor receptor (HER-2/neu) over-expression based on immunohistochemistry (IHC) (0 or 1+, 2+ if fluorescence in-situ hybridization [FISH] test is negative) or FISH (HER2/copy number of centromere of chromosome 17 [CEP17] ratio < 2.0 or < 4 Her-2/neu signals per nucleus)
* Any number of prior therapies for metastatic breast cancer is allowed; patients with weakly estrogen receptor positive breast cancer who received any number of endocrine agents for metastatic breast cancer will also be eligible
* Prior taxane is allowed (as long as the patient is not experiencing grade > 1 neuropathy and had no history of disease progression on a taxane therapy within 3 months prior to study enrollment)
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky >= 60%)
* Life expectancy of greater than 12 weeks
* Leukocytes >= 2,000/uL
* Absolute neutrophil count >= 1,500/uL
* Platelets >= 100,000/uL
* Total bilirubin less than or equal to the institution's upper limit of normal
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x institutional upper limit of normal (except for patients with liver metastases in whom AST/ALT can be < 5 x institutional upper limit of normal)
* Creatinine within normal institutional limits OR creatinine clearance >= 50 mL/min for patients with creatinine levels above institutional normal
* Left ventricular ejection fraction of > 50% on baseline echocardiography or multi-gated acquisition (MUGA) scan
* Corrected QT interval (QTc) of < 480 milliseconds
* Female subjects with child bearing potential must have a negative pregnancy test at screening; child bearing potential is defined as sexually active patients with menses less than 1 year prior to enrollment, < 65 years of age, have no history of oophorectomy or hysterectomy
* The effects of AT13387 on the developing human fetus are unknown; for this reason and because paclitaxel are known to be teratogenic; women of child-bearing potential and men must agree to use adequate contraception prior to study entry, for the duration of study participation and 3 months after completion of study treatment administration; adequate contraception includes methods such as oral contraceptives, double barrier method (condom plus spermicide or diaphragm), or abstaining from sexual intercourse; should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients who have had chemotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study
* Patients who are receiving any other investigational agents within 4 weeks or 5 half-lives (whichever is shorter) prior to the first dose of the study regimen
* Prior radiation therapy within 2 weeks prior to the first dose of the study regimen
* Patients in whom prior treatment related toxicities have not recovered to grade 1 or less (except for alopecia)
* Recent initiation of bone modifying therapy with a bisphosphonate or denosumab unless it has been started more than 4 weeks prior to the first dose of the study regimen; patients who are already enrolled in this study can initiate bone modifying therapy after the first set of re-staging scans (>= 8 weeks from cycle 1, day 1)
* Prior therapy with AT13387 or another HSP90 inhibitor
* Patients with known brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events; however, patients with previously treated and stable brain metastases are eligible as long as they are no longer requiring steroids, completed radiation therapy more than 2 weeks prior to the first dose of study regimen and have no seizures or worsening neurologic symptoms
* History of grade 3-4 immediate hypersensitivity reaction to paclitaxel
* History of clinically significant allergic reactions attributed to compounds of similar chemical or biologic composition to AT13387 or paclitaxel
* Based on investigator's brochure, AT13387 has no significant effects on inhibition or activation of cytochrome P450 (CYP), including 1A2, 3A4, 2D6, 2C9, and 2C19 at the half maximal inhibitory concentration (IC50) > 10 uM. Preclinical studies indicated that AT13387 is only a modest inhibitor of P-glycoprotein (P-gp). Paclitaxel is a substrate of CYP2C8 and CYP3A4. The use of CYP2C8 and CYP3A4 inhibitors/inducers while not prohibited in this study, is discouraged whenever feasible; concurrent use of strong CYP2C8 and CYP3A4 inhibitors/inducers should be documented and the principal investigator (PI) of the study shall be notified prior to dosing; as part of the enrollment/informed consent procedures, the patients will be counseled on the risk of interactions with other agents, and what to do if new medications need to be prescribed or if the patient is considering a new over-the-counter medicine or herbal product
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study because paclitaxel is a class D agent with the potential for teratogenic or abortifacient effects; because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with AT13387 and paclitaxel, breastfeeding should be discontinued if the mother is treated with AT13387 and paclitaxel
* Patients who are human immunodeficiency virus (HIV) positive on highly active anti-retroviral therapy (HAART) will be excluded from the study because of the potential for pharmacokinetic interactions with AT13387; in addition, these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy; appropriate studies will be undertaken in patients receiving combination antiretroviral therapy when indicated
* Inability to understand and sign informed consent
* Any other medical or psychiatric condition that in the opinion of the investigator would make the study therapy unsafe for the patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2016-01-15 (Actual); Primary Completion 2022-10-26 (Actual); Study Completion 2022-10-26 (Actual)

PRIMARY OUTCOMES:
Recommended phase 2 dose (R2PD) | Up to 28 days
  Defined as level at which no more than 1 of 6 patients experience a dose limiting toxicity (maximum tolerated dose or [MTD]); or doses of the combination below MTD, if in the opinion of the investigators, lower doses are better tolerated and safer.
Toxicity profile of onalespib in combination with paclitaxel | Up to 2 years
  Will be based on the Common Terminology Criteria for Adverse Events (CTCAE) version (v.)5.0.

SECONDARY OUTCOMES:
Pharmacokinetic (PK) parameters of onalespib | Pre-dose, immediately prior to end of infusion, 0.5, 1, 2, 4, 6, 8, and 24 hours after end of infusion on day -7 of course 1 and day 8 (and prior to starting paclitaxel, and immediately prior to end of infusion of paclitaxel on day 8)
  A descriptive analysis will be performed to define systemic exposure, drug clearance, and other pharmacokinetic parameters. The PK parameters will be summarized with simple summary statistics, including means, medians, ranges, and standard deviations (if numbers and distribution permit).
Pharmacokinetic (PK) parameters of paclitaxel | Pre-dose, immediately prior to end of infusion, 0.5, 1, 2, 4, 6, 8, and 24 hours after end of infusion on days 1 and 8 of course 1 (and immediately prior to end of infusion of onalespib, prior to starting paclitaxel on day 8)
  A descriptive analysis will be performed to define systemic exposure, drug clearance, and other pharmacokinetic parameters. The PK parameters will be summarized with simple summary statistics, including means, medians, ranges, and standard deviations (if numbers and distribution permit).
Overall response rate (partial response [PR]+ complete response [CR]) | Up to 6 months
  Will be assessed based on the Response Evaluation Criteria in Solid Tumors (RECIST) 1.1. Overall response will be assessed in all patients in an exploratory manner, using summary statistics, by dose level. Will also calculate corresponding 95% binomial confidence intervals for these response rates.
Response duration | From the time measurement criteria are met for complete response (CR) or partial response (PR) (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented, assessed up to 2 years
  Will be based on Response Evaluation Criteria in Solid Tumors (RECIST) 1.1.
Progression-free survival | From study enrollment to first documented disease progression according to Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 or death from any cause (whichever occurs first), assessed up to 2 years
  Progression free survival will be summarized using Kaplan and Meier methods, where patients who are event-free at the time of their last evaluation will be censored at that time point.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Wesolowski, Principal Investigator — Ohio State University Comprehensive Cancer Center LAO
Locations (4):
- United States (4):
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania

REFERENCES:
- [Derived] Williams NO, Quiroga D, Johnson C, Brufsky A, Chambers M, Bhattacharya S, Patterson M, Sardesai SD, Stover D, Lustberg M, Noonan AM, Cherian M, Bystry DM, Hill KL, Chen M, Phelps MA, Grever M, Stephens JA, Ramaswamy B, Carson WE 3rd, Wesolowski R. Phase Ib study of HSP90 inhibitor, onalespib (AT13387), in combination with paclitaxel in patients with advanced triple-negative breast cancer. Ther Adv Med Oncol. 2023 Dec 25;15:17588359231217976. doi: 10.1177/17588359231217976. eCollection 2023. PMID 38152697